CLINICAL TRIAL: NCT00966459
Title: Computed Tomography (CT) and Lung Function Data Collection for Computational Fluid Dynamics (CFD) in COPD Patients
Brief Title: Computed Tomography (CT) and Lung Function Data Collection for Computational Fluid Dynamics (CFD) in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Prof Dr Wilfried De Backer, University Hospital Antwerp, Department of Respiratory Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PML_DOC_0803
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Last update posted 2009-09-01 (Estimated); Status verified 2009-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Procedure: Computed Tomography

INTERVENTIONS:
Procedure: Computed Tomography — 1 low-dose CT is taken

SUMMARY:
In this study, 20 COPD patients will undergo a high-resolution/multi slice CT scan and lung function tests to obtain patient specific geometries of the central and peripheral small airways and patient specific boundary conditions.

With Computational Fluid Dynamics (CFD), the investigators will be able to reconstruct the geometry and measure the resistance of the peripheral airways.

In a later stage, CFD will be used to simulate the reaction of the airways on various inhalation medications.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with documented COPD based on the following criteria:

   * Smoking history of at least 10 pack-years.
   * Decreased Tiffeneau index (FEV1/(F)VC < 0.70).
2. Patients aged ≥ 40 years.
3. Patients should present moderate to very severe COPD with an FEV1 < 80% of predicted (GOLD 2, 3 and 4).
4. Patients should be treated according to GOLD guidelines.
5. Maintained on stable respiratory medications for 4 weeks prior to visit 1
6. Able to perform lung function tests.

Exclusion Criteria:

1. Patients below the age of 40.
2. Patients who are pregnant or are breast-feeding.
3. A respiratory infection or exacerbation of COPD in the four weeks prior to screening.
4. BMI > 35 kg/m².
5. Patients treated with BiPAP or CPAP.
6. Known active tuberculosis.
7. A history of asthma, cystic fibrosis, central bronchiectasis, interstitial lung disease or pulmonary thromboembolic disease.
8. A history of thoracotomy with pulmonary resection.
9. Active or untreated malignancy.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-11; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
To obtain patient specific geometries of the central and peripheral small airways
To obtain patient specific boundary conditions

SECONDARY OUTCOMES:
To measure the resistance of the peripheral airways
To measure the reaction of the airways on various inhalation medications

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Antwerp, Edegem, Antwerp, Belgium